CLINICAL TRIAL: NCT03696082
Title: A Precision Rehabilitation Approach to Counteract Age-Related Cognitive
Brief Title: A Precision Rehabilitation Approach to Counteract Age-Related Cognitive Declines
Acronym: CogEx
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding ended
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Fabrisia Ambrosio, Associate Professor, University of Pittsburgh
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Other
Other Study IDs: PRO17100528
Record Dates: First submitted 2018-09-13; First posted 2018-10-04 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Cognition Disorders; Brain Pathology; Physical Disability; Physical Activity; Aging
MeSH Terms: conditions — Cognition Disorders; Motor Activity | interventions — Exercise; Resistance Training; Yoga

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The outcome assessors will be masked to intervention assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Aerobic Activity (Experimental): Moderate-intensity exercise aerobic exercise that involves participating in activities similar to brisk walking that increase heart rate and breathing rate, with activity progressing to 150 minutes per week. Activities other than brisk walking, such as dance, aerobics, swimming, cycling or other activities that increase heart rate and breathing rate to a moderate intensity that can be sustained for at least 10 minutes will also be encouraged. This will require the participant to attend one supervised session each week for a period of 12 months with the remaining sessions being performed on their own without supervision.
  Interventions: Behavioral: Aerobic Activity
- Resistance Training (Experimental): Resistance exercise that involves participating in activities similar to lifting weights that cause the participant to work specific muscles of your body, with activity progressing to 150 minutes per week. This can involve using weight training machines, elastic tubes that create resistance, or weights such a dumbbells. This will require the participant to attend one supervised session each week for a period of 12 months with the remaining sessions being performed on their own without supervision.
  Interventions: Behavioral: Resistance Training
- Yoga (Experimental): Yoga involves a series of movements and poses that are performed in a specific sequence that are adapted to your ability, with activity progressing to 150 minutes per week. This will require the participant to attend one supervised session each week for a period of 12 months with the remaining sessions being performed on their own without supervision.
  Interventions: Behavioral: Yoga
- Health Education (Experimental): This involves the participant receiving information regarding aspects of health that are important for older adults, and also physical activity in the form of light stretching activities and movements. This will require the participant to attend one supervised session each week for a period of 12 months with the remaining sessions being performed on their own without supervision.
  Interventions: Behavioral: Health Education

INTERVENTIONS:
Behavioral: Aerobic Activity — Moderate-intensity exercise aerobic exercise that involves participating in activities similar to brisk walking that increase heart rate and breathing rate, with activity progressing to 150 minutes per week. Activities other than brisk walking, such as dance, aerobics, swimming, cycling or other activities that increase heart rate and breathing rate to a moderate intensity that can be sustained for at least 10 minutes will also be encouraged. This will require the participant to attend one supervised session each week for a period of 12 months with the remaining sessions being performed on their own without supervision.
  Arms: Aerobic Activity
Behavioral: Resistance Training — Resistance exercise that involves participating in activities similar to lifting weights that cause the participant to work specific muscles of your body, with activity progressing to 150 minutes per week. This can involve using weight training machines, elastic tubes that create resistance, or weights such a dumbbells. This will require the participant to attend one supervised session each week for a period of 12 months with the remaining sessions being performed on their own without supervision.
  Arms: Resistance Training
Behavioral: Yoga — Yoga involves a series of movements and poses that are performed in a specific sequence that are adapted to your ability, with activity progressing to 150 minutes per week. This will require the participant to attend one supervised session each week for a period of 12 months with the remaining sessions being performed on their own without supervision.
  Arms: Yoga
Behavioral: Health Education — This involves the participant receiving information regarding aspects of health that are important for older adults, and also physical activity in the form of light stretching activities and movements. This will require the participant to attend one supervised session each week for a period of 12 months with the remaining sessions being performed on their own without supervision.
  Arms: Health Education

SUMMARY:
This study examines the behavioral, molecular, and structural biomarkers of brain health that will allow for the stratification of individuals according to their "cognitive signature" and function. This study will randomize older adults into one of four interventions for a period of 12 months: 1) Aerobic Exercise, 2) Resistance Exercise, 3) Yoga Exercise, 4) Health Education (involves stretching and range of motion activities). This aims of this study will examine whether and how these different types of training interventions exert effects cognitive function, brain structure, biomarkers of brain health and cognition, and physical function.

DETAILED DESCRIPTION:
Physical activity is increasingly recognized to play a role in maintenance of brain health and attenuation of physical decline associated with aging. While physical activity has been shown to gradually decline with increasing age, initiation of an exercise protocol attenuates declines in cognition associated with advancing age, including impaired neurogenesis as well as decreased attention and learning. These benefits may be attributed, at least in part, to physical activity's role in maintaining an anti-inflammatory phenotype, and several clinical observational studies performed in older adults have shown an inverse relationship between self-reported physical activity and inflammatory biomarkers. Pre-clinical studies have also revealed that exposing aged animals to circulating factors derived from young animal counterparts significantly improves cognitive function and promotes neurogenesis.

A major limitation of clinical studies investigating the effect of physical activity on cognitive function is that subjects display considerable variability in their responses to the intervention. There are likely to be multiple biological pathways by which physical activity influences brain structure and function, and the type of physical activity that may be effective for influencing these pathways is likely to vary greatly. A better mechanistic understanding of how different modes of physical activity may target varying regions of the brain and other aspects of aging is therefore warranted.

This study examines the behavioral, molecular, and structural biomarkers of brain health that will allow for the stratification of individuals according to their "cognitive signature" and function. This study will randomize older adults into one of four interventions for a period of 12 months: 1) Aerobic Exercise, 2) Resistance Exercise, 3) Yoga Exercise, 4) Health Education (involves stretching and range of motion activities).

This aims of this study will examine whether and how these different types of training interventions exert differential effects on potential pathways of cognition and function in aged individuals, and the role of baseline subject characteristics in mediating these responses. The specific aims are:

1. To compare changes in cognitive function in response to three different types of physical activity (aerobic activity, resistance training activity, yoga) versus health education control.
2. To compare changes in brain structure in response to three different types of physical activity (aerobic activity, resistance training activity, yoga) versus health education control.
3. To compare biomarkers of brain health and cognition in response to three different types of physical activity (aerobic activity, resistance training activity, yoga) versus health education control.
4. To examine changes in physical function in response to three different types of physical activity (aerobic activity, resistance training activity, yoga) versus health education control.
5. To conduct post-hoc analyses to examine whether baseline measures of cognitive function, brain structure, biomarkers, or physical function influence responsiveness to any of the three different types of physical activity (aerobic activity, resistance training activity, yoga) versus health education control.

ELIGIBILITY:
Inclusion Criteria:

1. Age 65-80 years.
2. Sedentary, which is defined as regular participation over the past 3 months in <60 minutes per week of moderate-to-vigorous leisure-time or transportation-related physical activity performed in bouts of >10 minutes.
3. Independent ambulation without or with an cane or walking stick.
4. Able to walk (with or without assistive device such as a cane or walking stick) a distance of at least 400 meters based on self-report.
5. The ability to provide clearance from a physician for participation in the assessments and intervention aspects of this study.
6. Ability to provide informed consent.

Exclusion Criteria:

1. Reporting engaging in regular aerobic exercise, resistance exercise, or yoga exercise over the prior 3 months.
2. History of stroke, uncontrolled resting hypertension (systolic blood pressure ≥150 mmHg or diastolic blood pressure ≥100 mmHg), congestive heart failure, recent myocardial infarction, or other contraindications to engagement in moderate-intensity physical activity for at least 10 continuous minutes.
3. Incompatibility with the MRI environment (e.g. claustrophobia, metal implants, or body size, etc.)
4. Inability to attend the sessions as prescribed.
5. Consuming >1 alcoholic drink per day on >4 days per week, or current treatment for substance use disorder.
6. Report plans to relocate to a location not accessible to the study site or having employment, personal, or travel commitments that prohibit attendance to at least 80 percent of the scheduled intervention sessions and all of the scheduled assessments.
7. Use of a walker or rolling walker for ambulation.
8. SPPB score of <6 or unable to perform any of the 3 components of the total score [item score = 0].
9. Inability to complete the 400m walk test; or an unhealthy response to test [e.g., Systolic blood pressure >240 or diastolic blood pressure >115; or a drop in diastolic blood pressure > 10mm].
10. Depressive symptoms not controlled or treated.
11. List the medications that will exclude a participant (e.g., those that may complicate brain imaging, cognitive test, or biomarker testing or interpretation).
12. Degenerative neurological condition [e.g., Parkinson's Disease, multiple sclerosis].
13. Severe respiratory disease [eg COPD with shortness of breath], or use of supplemental oxygen.
14. Lower limb below or above knee amputation / prosthesis.
15. Score of <85 of the 3MS (Modified Mini-Mental State Exam).

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 78 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Brain Structure at 6 and 12 months | Baseline, 6 months, 12 months
  Measured used MRI and fMRI tasks.

SECONDARY OUTCOMES:
Change from Baseline Functional Fitness at 3, 6, and 12 months | Baseline, 3 months, 6 months, 12 months
  Assessed with the Short Physical Performance Battery
Change from Baseline Fitness at 3, 6, and 12 months | Baseline, 3 months, 6 months, 12 months
  Assessed with a 400 meter corridor walk.
Change from Baseline Repeatable Battery for the Assessment of Neuropsychological Status at 3, 6, and 12 months | Baseline, 3 months, 6 months, 12 months
  This is a brief standardized paper-and-pencil neurocognitive battery measuring immediate and delayed memory, attention, language, and visuospatial skills. The test comprises of 12 subtests that is administered by a trained examiner.
Change from Baseline Modified Mini-Mental Status Exam at 3, 6, and 12 months | Baseline, 3 months, 6 months, 12 months
  This is an expanded 100-point version of the original Mini-Mental Status Exam, administered in ~7 minutes, which assesses global cognitive function. This measure has very good reliability, validity, and sensitivity to moderate cognitive changes and has a proven record in clinical trials.
Change from Baseline Auditory Verbal Learning Test at 3, 6, and 12 months | Baseline, 3 months, 6 months, 12 months
  The participant is read a list of 15 words, 5 times. After each time, the participant is asked to immediately recall as many words as possible. Following the 5th recall, an interference list is presented, after which the participant is asked to spontaneously recall words from the original list. After a 10-minute interval has passed, the participant is asked again to recall as many words as possible from the original list.
Change from Baseline Physical Activity (minutes per week) at 3, 6, and 12 months | Baseline, 3 months, 6 months, 12 months
  Measured by Actigraphy
Change from Baseline Physical Activity (minutes per week) at 3, 6, and 12 months | Baseline, 3 months, 6 months, 12 months
  Measured by CHAMPS questionnaire.
Change from Baseline Physical Activity (minutes per week) at 3, 6, and 12 months | Baseline, 3 months, 6 months, 12 months
  Measured by Paffenbarger questionnaire.
Change from Baseline Sedentary Behavior (minutes per day) at 3, 6, and 12 months | Baseline, 3 months, 6 months, 12 months
  Measured by modified CARDIA questionnaire
Change from Baseline Sedentary Behavior (minutes per day) at 3, 6, and 12 months | Baseline, 3 months, 6 months, 12 months
  Measured by Actigraphy
Change from Baseline Peripheral biomarkers at 3, 6, and 12 months | Baseline, 3 months, 6 months, 12 months
  Assessed from venous blood collection and includes measures of neuroinflammation, neurogenesis, and cerebral vascularity

OTHER OUTCOMES:
Change from Baseline subjective well-being at 3, 6, and 12 months | Baseline, 3 months, 6 months, 12 months
  Measured by the Satisfaction with Life Scale (SWLS) 5-item questionnaire
Change from Baseline Mood at 3, 6, and 12 months | Baseline, 3 months, 6 months, 12 months
  Measured by the Positive and Negative Affect Schedule (PANAS) questionnaire
Change from Baseline Self-Efficacy for Physical Activity at 3, 6, and 12 months | Baseline, 3 months, 6 months, 12 months
  Measured by questionnaire with higher scores indicating greater self-efficacy
Change from Baseline Physical Activity Outcome Expectations at 3, 6, and 12 months | Baseline, 3 months, 6 months, 12 months
  Measured by questionnaire with higher scores indicating great outcome expectations.
Change from Baseline Physical Activity Barriers at 3, 6, and 12 months | Baseline, 3 months, 6 months, 12 months
  Measured by questionnaire with higher scores indicating greater barriers.
Change from Baseline Social Support for Physical Activity at 3, 6, and 12 months | Baseline, 3 months, 6 months, 12 months
  Measured by questionnaire with higher scores indicating greater social support
Change from Baseline Weight in kilograms at 3, 6, and 12 months | Baseline, 3 months, 6 months, 12 months
  Measured using a digital scale
Change from Baseline Height in centimeters at 3, 6, and 12 months | Baseline, 3 months, 6 months, 12 months
  Measured using a wall-mounted stadiometer
Change from Baseline resting systolic and diastolic blood pressure in mmHg at 3, 6, and 12 months | Baseline, 3 months, 6 months, 12 months
  Measured using an automated blood pressure system
Change from Baseline resting heart rate in beats per minute at 3, 6, and 12 months | Baseline, 3 months, 6 months, 12 months
  Measured using an automated system

CONTACTS AND LOCATIONS:
Overall Officials: John M. Jakicic, PhD, Principal Investigator — University of Pittsburgh; Fabrisia Ambrosio, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No